CLINICAL TRIAL: NCT02119988
Title: Transjugular Intrahepatic Portosystemic Shunt (TIPS) Using Covered Stents Combined With Variceal Embolization in the Prevention of Variceal Rebleeding for Patients With Cirrhosis : a Prospective, Open-labeled, Randomized, Controlled Trial
Brief Title: TIPS Combined With Variceal Embolization for the Prevention of Variceal Rebleeding in Patients With Cirrhosis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Air Force Military Medical University, China (Other)
Responsible Party: Principal Investigator, Guohong Han, M.D., Ph.D., Air Force Military Medical University, China
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: TIPS-Variceal embolization
Record Dates: First submitted 2014-04-17; First posted 2014-04-22 (Estimated); Last update posted 2022-10-25 (Actual); Status verified 2022-10

CONDITIONS: Liver Cirrhosis
Keywords: TIPS; Embolization; Variceal rebleeding
MeSH Terms: conditions — Liver Cirrhosis | interventions — Portasystemic Shunt, Transjugular Intrahepatic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- TIPS combined with variceal embolization (Experimental): The covered stents will be used for TIPS
  The gastroesophageal collaterals will be embolized during the procedure of TIPS
  Interventions: Procedure: TIPS; Procedure: Variceal Embolization
- TIPS alone (Active Comparator): The covered stents will be used for TIPS
  No embolization of any collateral will be performed during TIPS
  Interventions: Procedure: TIPS

INTERVENTIONS:
Procedure: TIPS — TIPS will be performed with a standard technique. TIPS revision will be planned if any evidence of shunt dysfunction is observed.
Procedure: Variceal Embolization — Embolization of gastroesophageal collaterals will be conducted via the same jugular vein before TIPS implantation. The major procedures includ (a) angiography of gastroesophageal collaterals after successful intrahepatic puncture of a branch of the portal vein and (b) embolization of gastroesophageal collaterals with coils of varying diameters, which result in the gastroesophageal collaterals disappearing at postembolization angiography.
  Arms: TIPS combined with variceal embolization

SUMMARY:
The purpose of this study is to determine whether TIPS combined with variceal embolization are effective in the prevention of variceal rebleeding in patients with liver cirrhosis.

DETAILED DESCRIPTION:
Variceal bleeding is one of the leading causes of death in patients with cirrhosis. Patients with cirrhosis surviving a variceal bleeding are at high risk of rebleeding (over 60% at 1 year), and mortality from each rebleeding episode is about 20%.

Placement of TIPS is a well-established technique that is highly effective in preventing recurrent variceal bleeding, especially if the TIPS is created with an expanded polytetrafluoroethylene (ePTFE)-covered stent, which has a significantly lower risk of shunt dysfunction than does TIPS created with bare stents. But the risk of hepatic encephalopathy greatly increases and the risk of recurrent variceal bleeding after TIPS placement remains an issue. Besides an insufficient decrease in portosystemic pressure gradient after TIPS creation alone, fragile variceal vessels also are considered a risk factor for recurrent bleeding.

Accordingly, TIPS combined with variceal embolization has been advocated to achieve the best result possible in preventing recurrent variceal bleeding. However, in recent American Association of the Study of Liver Disease (AASLD) practice guidelines and Baveno V consensus, no treatment strategies were clearly recommended maybe because the exact efficacy of this strategy remains unclear and high-quality randomized controlled trials still lacks.

So the investigators hypothesized that embolization of these collateral vessels may increase the blood flow within the shunt and into the liver, which can theoretically decrease the incidence of shunt dysfunction and encephalopathy, even can prolong the patients' survival.

ELIGIBILITY:
Inclusion Criteria:

* Signed written informed consent
* Dignosis of cirrhosis (clinical or by liver biopsy)
* Admission due to variceal bleeding occurred 5 to 42 days prior and standard treatment for secondary prophylaxis failed
* Age 18 to 75 years

Exclusion Criteria:

* Hepatic carcinoma and/or other malignancy diseases
* Portal vein thrombosis (≥50% of the lumen)
* Child-Pugh score>13 points
* Spontaneous recurrent hepatic encephalopathy
* Budd-Chiari syndrome
* Large spontaneous portosystemic shunts
* Sepsis
* Spontaneous bacterial peritonitis
* Uncontrollable hypertension
* Serious cardiac or pulmonary dysfunction
* Renal failure
* With TIPS contraindications
* Previous TIPS or collateral embolization,
* Pregnancy or breast-feeding
* History of organ transplantation

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 134 (Actual)
Dates: Start 2014-06-16 (Actual); Primary Completion 2020-11-20 (Actual); Study Completion 2020-11-20 (Actual)

PRIMARY OUTCOMES:
All-cause rebleeding | 2 years

SECONDARY OUTCOMES:
Variceal rebleeding | 2 years
Shunt dysfunction | 2 years
Hepatic encephalopathy | 2 years
Liver function changs | 2 years
Mortality | 2 years
Adverse events | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Guohong Han, PhD & MD, Principal Investigator — Xijing Hospital of Digestive Diseases, Fourth Military Medical University
Locations (2):
- China (2):
  - Xijing Hospital of digestive disease, Fourth Military Medical University, Xi'an, Shaanxi
  - Xijing Hospital of Digestive Diseases, Fourth Military Medical University, Xi'an, Shaanxi

REFERENCES:
- [Derived] Lv Y, Chen H, Luo B, Bai W, Li K, Wang Z, Xia D, Guo W, Wang Q, Li X, Yuan J, Cai H, Xia J, Yin Z, Fan D, Han G. Transjugular intrahepatic portosystemic shunt with or without gastro-oesophageal variceal embolisation for the prevention of variceal rebleeding: a randomised controlled trial. Lancet Gastroenterol Hepatol. 2022 Aug;7(8):736-746. doi: 10.1016/S2468-1253(22)00087-5. Epub 2022 May 17. PMID 35588750